CLINICAL TRIAL: NCT04070105
Title: No Power Bionic Lower Extremity Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Deanna H Gates, Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00150407
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Amputation; Amputation, Traumatic; Amputation; Traumatic, Leg, Lower
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will walk with their standard prosthesis, a commercial high activity foot, and then the new design of CAESAR foot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- CAESAR Foot, Prescribed Feet, AllPro (Experimental): Participants will walk and run with different prostheses on different days in a laboratory. The order of testing is CAESAR Foot, Prescribed Feet, AllPro.
  Interventions: Device: Compliant Adaptive Energy Storage and Return Foot; Device: AllPro
- CAESAR Foot, AllPro, Prescribed Feet (Experimental): Participants will walk and run with different prostheses on different days in a laboratory. The order of testing is CAESAR Foot, AllPro, Prescribed Feet
  Interventions: Device: Compliant Adaptive Energy Storage and Return Foot; Device: AllPro
- Prescribed Feet, AllPro, CAESAR Foot (Experimental): Participants will walk and run with different prostheses on different days in a laboratory. The order of testing is Prescribed Feet, AllPro, CAESAR Foot
  Interventions: Device: Compliant Adaptive Energy Storage and Return Foot; Device: AllPro
- Prescribed Feet, CAESAR Foot, AllPro (Experimental): Participants will walk and run with different prostheses on different days in a laboratory. The order of testing is Prescribed Feet, CAESAR Foot, AllPro
  Interventions: Device: Compliant Adaptive Energy Storage and Return Foot; Device: AllPro
- AllPro, Prescribed Feet, CAESAR Foot (Experimental): Participants will walk and run with different prostheses on different days in a laboratory. The order of testing is AllPro, Prescribed Feet, CAESAR Foot
  Interventions: Device: Compliant Adaptive Energy Storage and Return Foot; Device: AllPro
- AllPro, CAESAR Foot, Prescribed Feet, (Experimental): Participants will walk and run with different prostheses on different days in a laboratory. The order of testing is AllPro, CAESAR Foot, Prescribed Feet
  Interventions: Device: Compliant Adaptive Energy Storage and Return Foot; Device: AllPro

INTERVENTIONS:
Device: Compliant Adaptive Energy Storage and Return Foot — The primary concept of the CAESAR foot is to switch from a walking foot to a running foot with the push of a button
  Other Names: CAESAR Foot
Device: AllPro — Participants will be fit with a high activity foot designed to be used for walking and running

SUMMARY:
Typically people need separate prosthetic feet for running and walking. To bridge the gap, this study will test the Compliant Adaptive Energy Storage and Return (CAESAR) foot. This foot can change from a walk mode to a run mode with the push of a button. The investigators will test and improve this foot design mechanically, and then test this design on individuals with lower limb amputation in a lab setting. The goal of this project is to develop a passive prosthetic foot that can serve two purposes in someone's daily life: walking and running, to allow them to be more active.

DETAILED DESCRIPTION:
Typically people need separate prosthetic feet for running and walking. To bridge the gap, this study will test the Compliant Adaptive Energy Storage and Return (CAESAR) foot. This foot can change from a walk mode to a run mode with the push of a button. The investigators will test and improve this foot design mechanically, and then test this design on individuals with lower limb amputation in a lab setting. The goal of this project is to develop a passive prosthetic foot that can serve two purposes in someone's daily life: walking and running, to allow them to be more active. Here we will test this device to determine how it affects the user's mechanics during running and walking. Participants will come to a research laboratory for three test sessions where they will run and walk in their current foot, a commercial high-activity foot, and the prototype CAESAR foot.

ELIGIBILITY:
Patient Population:

Inclusion Criteria:

* At least 18 years old
* Transtibial amputation of one or both legs
* Classified as K3 or K4 on the Medicare Functional Classification Level
* Use of a well-fitting prosthetic socket and prosthetic foot for at least 6 months
* Able to walk and run without assistance

Exclusion Criteria:

* Significant injury to intact limb
* History of balance impairments or neurologic disorders
* Significant cardiovascular or respiratory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants enrolled in the study and tested a prototype foot to assess stiffness. A foot was then manufactured for them specifically. Due to COVID19 pauses in collection there was a significant gap between manufacturing the prosthetic feet and human subjects testing. One participant was no longer available to complete laboratory testing. The order of testing was randomized between participants, such that all participants completed testing in a different order.
Groups:
- CAESAR, Then Prescribed, Then AllPro; CAESAR, Then AllPro, Then Prescribed; Prescribed, Then AllPro, Then CAESAR; Prescribed, Then CAESAR, Then AllPro; AllPro, Then CAESAR, Then Prescribed; AllPro, Then Prescribed, Then CAESAR: Participants will walk and run with three prostheses in random order
Period: Overall Study
Arm/Group | CAESAR, Then Prescribed, Then AllPro | CAESAR, Then AllPro, Then Prescribed | Prescribed, Then AllPro, Then CAESAR | Prescribed, Then CAESAR, Then AllPro | AllPro, Then CAESAR, Then Prescribed | AllPro, Then Prescribed, Then CAESAR
Started | 0 | 2 | 1 | 1 | 1 | 1
Completed | 0 | 2 | 1 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Prosthetic Foot Intervention: Participants will walk and run with one of three different prostheses, their standard of care running and walking prostheses, a new prosthesis designed to switch orientation of the foot with a push of a button, and a high activity foot (AllPro, Fillauer, Chattanooga, TN)
  Compliant Adaptive Energy Storage and Return Foot: The primary concept of the CAESAR foot is to switch from a walking foot to a running foot with the push of a button
  Conventional Prosthetic Foot: This is a commercial prosthetic foot that has been prescribed to the individual
  Commercial High Activity Foot: This is a commercially available prosthetic foot designed for high-activity individuals
Arm/Group | Prosthetic Foot Intervention
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6
Height (m) [Mean (Standard Deviation); unit: meters] | 1.75 (0.10)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 80.0 (8.3)

OUTCOME MEASURES:

1. Primary Outcome: Peak Propulsive Ground Reaction Force on the Prosthetic Side During Walking
Description: Participants will walk over sensors that measure the force under their foot. Peak ground reaction force in the anterior direction is measured in Newtons and then divided by the individual's body weight (BW). The resultant force is measured in Body-weights.
Time Frame: All conditions were complete during 3 lab visits, approximately four hours long
Population: Participants walked with each of three feet: prescribed, CAESAR, and AllPro
Measure: Mean (Standard Deviation); unit: Body-weights
Groups:
- Prescribed: This is a commercial prosthetic foot that has been prescribed to the individual
- AllPro: This is a commercially available prosthetic foot designed for high-activity individuals
- CAESAR: Compliant Adaptive Energy Storage and Return Foot: The primary concept of the CAESAR foot is to switch from a walking foot to a running foot with the push of a button
Arm/Group | Prescribed | AllPro | CAESAR
Number analyzed (Participants) | 5 | 5 | 5
Body-weights | .175 (0.043) | .166 (0.022) | .166 (0.013)

2. Primary Outcome: Participants Perceived Comfort When Using Different Prosthetic Feet During Walking
Description: Participants were asked their perceived comfort on a visual analog scale from 0 (most uncomfortable) to 100 (most comfortable)
Time Frame: All conditions were complete during 3 lab visits, approximately four hours long
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prescribed | AllPro | CAESAR
Number analyzed (Participants) | 5 | 5 | 5
score on a scale | 84.8 (11.1) | 80.6 (18.7) | 77.4 (23.9)

3. Primary Outcome: Peak Propulsive Ground Reaction Force on the Prosthetic Side During Running
Description: Participants will run on a treadmill with force sensors below the treadmill belt. Data will be measured in Newtons and then normalized by dividing by body weight.
Time Frame: All conditions were complete during 3 lab visits, approximately four hours long
Population: Participants ran with each of three feet: prescribed, CAESAR, and AllPro
Measure: Mean (Standard Deviation); unit: Body-weights
Groups:
- Prescribed: This is a commercial prosthetic foot that has been prescribed to the individual that they used for running. For some individuals this was a running foot, while for others it was not
Arm/Group | Prescribed | AllPro | CAESAR
Number analyzed (Participants) | 3 | 2 | 3
Body-weights | 0.093 (0.006178) | 0.079 (0.005169) | .154 (0.004942)

4. Secondary Outcome: Net V02 (Metabolic Cost) During Running
Description: Participants will wear a mask that measures their rate of oxygen consumption while they run for 5 minutes at a comfortable pace
Time Frame: All conditions were complete during 3 lab visits, approximately four hours long
Population: Participants who could run comfortably on the treadmill for 5 minutes with that foot
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Prescribed | AllPro | CAESAR
Number analyzed (Participants) | 3 | 2 | 3
mL/kg/min | 25.66 (2.93) | 26.86 (2.99) | 27.68 (2.52)

5. Primary Outcome: Participants Perceived Comfort When Using Different Prosthetic Feet During Running
Description: as for outcome 2
Time Frame: All conditions were complete during 3 lab visits, approximately four hours long
Population: Participants who ran in the lab with each foot style. One participant did not complete the survey with his prescribed foot
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prescribed | AllPro | CAESAR
Number analyzed (Participants) | 4 | 5 | 5
score on a scale | 51.8 (27.2) | 59.6 (23.3) | 66.4 (36.5)

ADVERSE EVENTS:
Time Frame: During each of the three, approximately 4 hour, data collection sessions
Arm/Group | Prosthetic Foot Intervention
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Six participants were enrolled and we built six feet for those individuals. Due to delays because of COVID pauses in human subjects testing, only five were available to test the final foot design. Of these, only three were able to run on a treadmill comfortably for five minutes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT04070105/Prot_SAP_000.pdf